CLINICAL TRIAL: NCT04946201
Title: The Effect of Upper Premolars Extraction on Obstructive Sleep Apnea in Growing Children With Prominent Upper Front Teeth
Brief Title: Premolar Extractions for Obstructive Sleep Apnea in Children With Overjet
Status: Suspended | Type: Observational
Why Stopped: Reduction in staff
Sponsor: Mohamed Bazina (Other)
Responsible Party: Sponsor-Investigator, Mohamed Bazina, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 63668
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea; Malocclusion
Keywords: orthodontic; braces; extraction; teeth; overjet
MeSH Terms: conditions — Sleep Apnea, Obstructive; Malocclusion; Overbite

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Extractions: Patients in this group will undergo dental extractions.
- Without Extractions: Patients in this group will not undergo dental extractions.

SUMMARY:
This research aims to provide pediatric patients with polysomnography (a sleep study) before and after orthodontic treatment to determine if the extraction of upper premolars for treating excessive overjet results in an increase of the AHI (Apnea Hypopnea Index) compared to similar patients treated without upper premolar extractions.

ELIGIBILITY:
Inclusion Criteria:

* 10-15 years old
* registered orthodontic patients
* able to undergo routine orthodontic care and are registered to obtain an orthodontic appliance in the future.
* do not have a high care need
* no known hypercapnia or hypoventilation
* no known allergies or nose blockages
* diagnosed as Class II Division I (=6mm of overjet) and bilateral Class II half cusp or unilateral Class II full cusp.

Exclusion Criteria:

* known hypercapnia or hypoventilation
* patients with hypertrophic tonsils and adenoids
* patients with allergies or nose blockages that interfere with breathing
* patients who are not registered as orthodontic patients at research sites deemed acceptable to undergo routine orthodontic care

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Registered orthodontic patients at the College of Dentistry and Turfland Dental Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Risk of Obstructive Sleep Apnea | 30 months
  Percentage of participants who develop obstructive sleep apnea following orthodontic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Bazina, DDS, MSD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No